CLINICAL TRIAL: NCT00523575
Title: Effectiveness and Cost-effectiveness of Nutritional Screening and Intervention in Elderly Subjects After Hip Fracture
Brief Title: Nutritional Intervention in Hip Fracture Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: PC Dagnelie, PhD, Maastricht University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 06-3-098; ZonMw 80-007022-98-07510
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Hip Fracture; Malnutrition
Keywords: Elderly; Osteoporosis; hip fracture; malnutrition; nutritional support
MeSH Terms: conditions — Hip Fractures; Malnutrition; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- C (No Intervention): Usual nurse and dietetic care
- I (Experimental): Intensive nutritional support composed of oral dietary supplement combined with dietetic counselling.
  Interventions: Dietary Supplement: Cubitan

INTERVENTIONS:
Dietary Supplement: Cubitan — 400 ml/d
  Other Names: Nutricia: Cubitan
  Arms: I

SUMMARY:
Hip fractures are highly prevalent and are expected to increase due to the ageing population. Malnutrition is often present in these patients and is associated with prolonged convalescence, lower mobility, lower mental function, lower quality of life and higher complication rate. Nutritional intervention starting soon after hospital admission might reduce complication rate and total length-of-stay by improving nutritional and functional status. Research questions are:

1. Does nutritional intervention reduce total length-of-stay?
2. Is nutritional intervention cost-effective?
3. Can nutritional screening contribute to targeting of nutritional intervention, and thereby reduce costs without loss of effectiveness?

Patients randomized to the intervention group will receive oral nutritional supplements (protein and energy enriched) and regular dietetic counselling during hospitalisation and after discharge at patients' homes for 3 months. Patients in the control group will receive usual nurse and dietetic care. Outcome measurements will be taken at baseline, 3 months and 6 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Admission to one of the participating hospitals because of a proximal femur fracture
* Age 55 years and older

Exclusion Criteria:

* Periprosthetic or pathologic fracture
* Diseases of bone metabolism, e.g. Paget, primary/secondary bone tumors, hyperparathyroidism, M. Kahler
* Life expectation of less than one year due to underlying disease (e.g. cancer)
* Presence of dementia or other severely impaired cognitive function
* Inability to communicate in Dutch language
* Nutritional intervention prior to admission
* Patients who are bedridden
* Patients who are too ill or for any other reason not able to participate adequately in follow-up

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Total length of hospital stay and rehabilitation clinics | baseline, 3 months and 6 months after inclusion

SECONDARY OUTCOMES:
Nutritional status, hip functionality, physical disability, fatigue, quality of life. | baseline, 3 months and 6 months after inclusion
Cost questionnaire, informal care questionnaire. | baseline, 3 months and 6 months after inclusion
Rate of complications | baseline, 3 months and 6 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: P C Dagnelie, PhD, Principal Investigator — Maastricht University - Faculty of Health Medicine and Life Sciences - Department of Epidemiologie; P LM Reijven, PhD, Principal Investigator — Maastricht University Hospital - Department of Dietetics & Maastricht University - Faculty of Health Medicine and Life Sciences - Department of Epidemiology
Locations (3):
- Netherlands (3):
  - Atrium MC, Heerlen
  - Maastricht University Hospital, Maastricht
  - Maaslandziekenhuis, Sittard

REFERENCES:
- [Derived] Wyers CE, Reijven PLM, Breedveld-Peters JJL, Denissen KFM, Schotanus MGM, van Dongen MCJM, Eussen SJPM, Heyligers IC, van den Brandt PA, Willems PC, van Helden S, Dagnelie PC. Efficacy of Nutritional Intervention in Elderly After Hip Fracture: A Multicenter Randomized Controlled Trial. J Gerontol A Biol Sci Med Sci. 2018 Sep 11;73(10):1429-1437. doi: 10.1093/gerona/gly030. PMID 30204859
- [Derived] Breedveld-Peters JJ, Reijven PL, Wyers CE, van Helden S, Arts JJ, Meesters B, Prins MH, van der Weijden T, Dagnelie PC. Integrated nutritional intervention in the elderly after hip fracture. A process evaluation. Clin Nutr. 2012 Apr;31(2):199-205. doi: 10.1016/j.clnu.2011.10.004. Epub 2011 Oct 28. PMID 22035956
- [Derived] Wyers CE, Breedveld-Peters JJ, Reijven PL, van Helden S, Guldemond NA, Severens JL, Verburg AD, Meesters B, van Rhijn LW, Dagnelie PC. Efficacy and cost-effectiveness of nutritional intervention in elderly after hip fracture: design of a randomized controlled trial. BMC Public Health. 2010 Apr 27;10:212. doi: 10.1186/1471-2458-10-212. PMID 20423469